CLINICAL TRIAL: NCT03195400
Title: Pathogenesis of Youth Onset Type 2 Diabetes and Prediabetes
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000020183; 1R01DK111038-01A1 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-06-22 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: IGT - Impaired Glucose Tolerance; T2D
MeSH Terms: conditions — Glucose Intolerance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from whole blood with the use of a Flexigene Kit (Qiagen) and genotyping will be performed using a matrix assisted based laser desorption-ionization time of flight mass spectrometry on the MassARRAY platform (Sequenom). DNA sample is obtained with fasting samples during the OGTT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CC Genotype: Subjects who have not already been tested previously will be tested for the TCF7L2 genotype to determine if they are TT or CC. An anticipated 50 obese CC adolescents with IGT or pre-IGT with similar age, pubertal stage, ethnicity and Body Mass Index (BMI) will enrolled. Subjects will undergo Oral Glucose Tolerance Test, Hyperglycemic Clamp, Isoglycemic Intravenous Glucose Test IsoG IVGT and Hyperinsulinemic Euglycemic Clamp and 2H20.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Diagnostic Test: Hyperglycemic Clamp; Diagnostic Test: Isoglycemic Intravenous Glucose Test; Diagnostic Test: Hyperinsulinemic Euglycemic Clamp and 2H20
- TT Genotype: Subjects who have not already been tested previously will be tested for the TCF7L2 genotype to determine if they are TT or CC. An anticipated 50 TT subjects will be enrolled in this group. An anticipated 50 obese TT adolescents with IGT or pre-IGT with similar age, pubertal stage, ethnicity and Body Mass Index (BMI) will be enrolled. Subjects will undergo Oral Glucose Tolerance Test, Hyperglycemic Clamp, Isoglycemic Intravenous Glucose Test IsoG IVGT and Hyperinsulinemic Euglycemic Clamp and 2H20
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Diagnostic Test: Hyperglycemic Clamp; Diagnostic Test: Isoglycemic Intravenous Glucose Test; Diagnostic Test: Hyperinsulinemic Euglycemic Clamp and 2H20

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — The oral glucose tolerance test (OGTT) measures the body's ability to use a type of sugar, called glucose, that is the body's main source of energy. An OGTT can be used to diagnose prediabetes and diabetes.
  Other Names: OGTT
Diagnostic Test: Hyperglycemic Clamp — Test of beta-cell function and insulin secretion. Involves increasing and maintaining blood glucose concentration with IV variable infusion of dextrose.
  Other Names: Infusion Study
Diagnostic Test: Isoglycemic Intravenous Glucose Test — Test which exposes pancreas to blood glucose levels matched to the ones obtained at the OGTT.
  Other Names: IsoG IVGT
Diagnostic Test: Hyperinsulinemic Euglycemic Clamp and 2H20 — Test is used to assess insulin effects on hepatic glucose production.
  Other Names: E Clamp with labeled water

SUMMARY:
Type 2 Diabetes (T2D) in obese youth is often preceded by a prediabetic state called: Impaired Glucose Tolerance (IGT), which is associated with a pre-existing defect in insulin secretion. This study intends to determine if genetic factors are associated with defects in insulin secretion, the incretin system and hepatic insulin resistance in obese adolescents. The long-term goal of this study is to generate information on both the genetics as well as the pathophysiology of Type 2 Diabetes in Youth, which ultimately might guide the investigators towards better preventive and treatment avenues.

DETAILED DESCRIPTION:
The Specific Aims of this study are:

Aim 1a. To delineate the effects of TCF7L2 rs7903146 on functional Beta-Cell Capacity in obese adolescents with Impaired Glucose Tolerance (IGT) and pre-IGT.

Aim 1b. To determine if the risk genotype in TCF7L2 is associated with worsening in beta cell function longitudinally, thereby affecting changes in glucose tolerance.

Aim 2. To examine the functional effect of the rs7903146 variant in the TCF7L2 gene on a) incretin effect in obese adolescents with IGT and pre-IGT.

Aim 3. To determine the functional effects of TCF7L2 rs7903146 SNP on hepatic glucose fluxes in obese adolescents with IGT and pre-IGT.

ELIGIBILITY:
Inclusion Criteria:

* Good general health, taking no medication on a chronic basis;
* Age 12 to 18 yrs, in puberty (girls and boys: Tanner stage II - IV),
* BMI (BMI >85th%) indicating obesity,
* Girls who are menstruating must have a negative pregnancy test during the study and, when possible, be in the follicular phase during infusion study visits (The follicular phase will be identified according to the last menstrual period record and/or according to the oral contraceptive assumption schedule. The investigators will not perform ovulation testing or hormonal assays);
* Subject must have normal liver and kidney function, amylase and lipase levels.
* Pre-IGT or IGT
* TT or CC genotype.

Exclusion Criteria:

* Baseline creatinine >1.0 mg;
* Pregnancy;
* Presence of endocrinopathies (e.g. Cushing syndrome);
* Cardiac, renal or pulmonary or other chronic illness;
* Adolescents with psychiatric disorder or with substance abuse history and taking the drugs that affect glucose metabolism, such as any form of steroids, antipsychotics, progesterone preparations, and others.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be selected from the Yale Pediatric Obesity Clinic or from the existing cohort of subjects who have had Oral Glucose Tolerance Tests and genotyping. Subjects will be Pre IGT and IGT adolescents 12-18 years old with either the CC or TT genotype. 50 CC pre IGT/IGT obese patients and 50 TT pre IGT/IGT obese patients will be rectruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance status | Baseline
  An oral glucose tolerance test will be performed to assess glucose tolerance status to determine if subjects are pre-IGT or IGT
Genotype | Baseline
  DNA screening to measure whether subject is CC or TT genotype
Beta cell capacity | Baseline
  AIRmax stimulation test during the hyperglycemic clamp to ascertain the maximal acute insulin response (AIR) to arginine, which is a measure of functional beta cell capacity.
Incretin effect | 3weeks to 1 month post Baseline testing
  Subjects will undergo the IsoIVGT test with GLP-1 measurements to measure the incretin effect
Beta cell function (longitudinally) | 2 years post Baseline
  The AIRmax stimulation test during the hyperglycemic clamp will be repeated at 2 years to determine if genotype TCF7L2 contributes to worsening in beta cell function longitudinally
Hepatic glucose fluxes | 2 months post baseline testing
  Measurements from the Hyperinsulinemic Euglycemic Clamp/ 2H20 Study will be used to assess insulin effects on hepatic glucose production and glycerol kinetics isotopes and the deuterium enrichment at carbons 2 and 5 (C2 and C5) of plasma glucose providing information on glucose fluxes

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided